CLINICAL TRIAL: NCT06455150
Title: Prevalence of Pelvic Floor Dysfunctions in Female Badminton Athletes and Sedentary: Protocol of an Observational Case-Control Study
Brief Title: Prevalence of Pelvic Floor Dysfunctions in Female Badminton Athletes and Sedentary
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Lara Díaz Álvarez, Physiotherapist, University of Alcala
Other Study IDs: CEIM/2024/2/030
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Pelvic Floor Disorders
Keywords: prevalence; pelvic floor disorders; racquet sports; sedentary behavior; women
MeSH Terms: conditions — Pelvic Floor Disorders; Sedentary Behavior | interventions — Singing; Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Female badminton athletes
  Interventions: Other: Assessment of pelvic floor dysfunctions' symptoms and sings, pelvic floor muscle strength and quality of life
- Controls: Sedentary women
  Interventions: Other: Assessment of pelvic floor dysfunctions' symptoms and sings, pelvic floor muscle strength and quality of life

INTERVENTIONS:
Other: Assessment of pelvic floor dysfunctions' symptoms and sings, pelvic floor muscle strength and quality of life — It will be assessed the presence of urinary incontinence, anal incontinence, pelvic organ prolapse and female sexual dysfunction' symptoms by using the questionaries validated to Spanish population "International Consultation on Incontinence Questionnaire-Short Form", "Pelvic Floor Distress Inventory Short Form" and "Female Sexual Function Index"; in addition, the sign of stress urinary incontinence and pelvic organ prolapse will be assessed by using the cough stress test and Pelvic Organ Prolapse Quantification System, the pelvic floor muscle strength by using manometry, and quality of life by using SF-12 questionnaire.

SUMMARY:
The objective of the study is to know the prevalence of pelvic floor dysfunctions in female badminton athletes compared to sedentary women, and the hypothesis is that the prevalence of pelvic floor dysfunctions is going to be higher in female badminton athletes.

DETAILED DESCRIPTION:
After being informed about the study, all participants giving written informed consent will complete the personal data questionnaire and the questionnaires validated to Spanish population "International Consultation on Incontinence Questionnaire-Short Form" (ICIQ-SF), "Pelvic Floor Distress Inventory Short Form" (PFDI-20), "Female Sexual Function Index" (FSFI) and the SF-12 questionnaire. After that, inclusion and exclusion criteria will be assessed, and participants will be allocated into cases and controls group. Both groups will undergo the same procedures. Firstly, the evaluation of stress urinary incontinence and pelvic organ prolapse signs will be performed by using the cough stress test and Pelvic Organ Prolapse Quantification System; and secondly, the evaluation of pelvic floor muscle strength by using manometry.

ELIGIBILITY:
Inclusion Criteria:

* Cases: women who practice recreational badminton and/or are federated and compete.
* Controls: sedentary women and/or do not meet the recommendations of the World Health Organization (150-300 minutes of moderate-intensity aerobic physical activity or 75-150 minutes of vigorous-intensity aerobic physical activity).

Exclusion Criteria:

* Connective tissue diseases (Ehlers-Danlos syndrome, Marfan syndrome or hypermobility syndrome).
* Pregnant at the time of the study.
* Give birth in the last 12 months.
* Not understanding Spanish language.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women from Comunidad de Madrid (Spain) who want to participate and fullfil the inclusion criteria.
  In the cases group, women from badminton clubs register at the "Federación Madrileña de Bádminton" and University clubs or not register in this federation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence symptoms | 1 assessment when participants are recruited
  International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF): total score greater than 0 is positive for urinary incontinence
Anal incontinence and pelvic organ prolapse symptoms | 1 assessment when participants are recruited
  Pelvic Floor Distress Inventory Short Form (PFDI-20): item 3 pelvic organ prolapse symptom, item 9 solid fecal incontinence symptom, item 10 liquid fecal incontinence symptom, item 11 flatal incontinence symptom, item 13 fecal (rectal) urgency symptom. Affirmative answer is positive for the symptoms.
Female sexual dysfunction symptoms | 1 assessment when participants are recruited
  Female Sexual Function Index (FSFI): total score less or equal to 26 points is positive for female sexual dysfunction risk

SECONDARY OUTCOMES:
Stress urinary incontinence sign | 1 assessment when participants are recruited
  Cough stress test: with a comfortable sensation of a full bladder (200-400 mL), it is considered positive when a leakage of urine is visualized at the urethral meatus at the same time as coughing (between 1 and 4 repetitions). If the result is negative, the test should be repeated in a standing position (accessory test).
Pelvic organ prolapse sign | 1 assessment when participants are recruited
  Pelvic Organ Prolapse Quantification System: the patient with empty bladder and rectum (if possible), the presence, type and stage of pelvic organ prolapse will be assessed by a gynecologist.
Pelvic floor muscle strength | 1 assessment when participants are recruited
  Manometry: probe will be inserted, calibrated to 0 and asked to perform 3 maximum voluntary contractions of the pelvic floor muscle, 10 seconds break in between, after the verbal instruction "squeeze and lift the probe as strongly as possible". The total score will be the average of the three values. Measured in centimetres of water.
Participant's quality of life | 1 assessment when participants are recruited
  SF-12 questionnaire: total score greater than 50 points, better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Lara Díaz Álvarez, Principal Investigator
Locations (1):
- Faculty of Nursing and Physiotherapy of the University of Alcala, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eickmeyer SM. Anatomy and Physiology of the Pelvic Floor. Phys Med Rehabil Clin N Am. 2017 Aug;28(3):455-460. doi: 10.1016/j.pmr.2017.03.003. Epub 2017 May 27. PMID 28676358
- [Background] Donnelly GM, Moore IS. Sports Medicine and the Pelvic Floor. Curr Sports Med Rep. 2023 Mar 1;22(3):82-90. doi: 10.1249/JSR.0000000000001045. PMID 36866951
- [Background] Torres Lacomba M, Navarro Brazález B, Arranz Martín B. Fisioterapia y suelo pélvico: condiciones específicas en la vida de la mujer. Fisioterapia del Suelo Pélvico. Manual para la prevención y el tratamiento en la mujer, en el hombre y en la infancia. Madrid: Editorial Médica Panamericana; 2022. p. 145-60. ISBN: 978-84-9110-453-7.
- [Background] Cabello Manrique D, Gonzalez-Badillo JJ. Analysis of the characteristics of competitive badminton. Br J Sports Med. 2003 Feb;37(1):62-6. doi: 10.1136/bjsm.37.1.62. PMID 12547746
- [Background] Giagio S, Salvioli S, Pillastrini P, Innocenti T. Sport and pelvic floor dysfunction in male and female athletes: A scoping review. Neurourol Urodyn. 2021 Jan;40(1):55-64. doi: 10.1002/nau.24564. Epub 2020 Nov 2. PMID 33137211
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. doi: 10.1016/j.jclinepi.2007.11.008. PMID 18313558
- [Background] Peinado-Molina RA, Hernandez-Martinez A, Martinez-Vazquez S, Rodriguez-Almagro J, Martinez-Galiano JM. Pelvic floor dysfunction: prevalence and associated factors. BMC Public Health. 2023 Oct 14;23(1):2005. doi: 10.1186/s12889-023-16901-3. PMID 37838661
- [Background] Teixeira RV, Colla C, Sbruzzi G, Mallmann A, Paiva LL. Prevalence of urinary incontinence in female athletes: a systematic review with meta-analysis. Int Urogynecol J. 2018 Dec;29(12):1717-1725. doi: 10.1007/s00192-018-3651-1. Epub 2018 Apr 13. PMID 29654349
- [Background] Sánchez Sánchez B. Epidemiología y factores de riesgo en las disfunciones del suelo pélvico. Fisioterapia del Suelo Pélvico. Manual para la prevención y el tratamiento en la mujer, en el hombre y en la infancia. Madrid: Editorial Médica Panamericana; 2022. p. 101-7. ISBN: 978-84-9110-453-7.
- [Background] Tim S, Mazur-Bialy AI. The Most Common Functional Disorders and Factors Affecting Female Pelvic Floor. Life (Basel). 2021 Dec 14;11(12):1397. doi: 10.3390/life11121397. PMID 34947928
- [Background] Espuna Pons M, Rebollo Alvarez P, Puig Clota M. [Validation of the Spanish version of the International Consultation on Incontinence Questionnaire-Short Form. A questionnaire for assessing the urinary incontinence]. Med Clin (Barc). 2004 Mar 6;122(8):288-92. doi: 10.1016/s0025-7753(04)74212-8. Spanish. PMID 15030739
- [Background] Sanchez-Sanchez B, Torres-Lacomba M, Yuste-Sanchez MJ, Navarro-Brazalez B, Pacheco-da-Costa S, Gutierrez-Ortega C, Zapico-Goni A. Cultural adaptation and validation of the Pelvic Floor Distress Inventory short form (PFDI-20) and Pelvic Floor Impact Questionnaire short form (PFIQ-7) Spanish versions. Eur J Obstet Gynecol Reprod Biol. 2013 Sep;170(1):281-5. doi: 10.1016/j.ejogrb.2013.07.006. Epub 2013 Jul 25. PMID 23891390
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Sanchez-Sanchez B, Navarro-Brazalez B, Arranz-Martin B, Sanchez-Mendez O, de la Rosa-Diaz I, Torres-Lacomba M. The Female Sexual Function Index: Transculturally Adaptation and Psychometric Validation in Spanish Women. Int J Environ Res Public Health. 2020 Feb 5;17(3):994. doi: 10.3390/ijerph17030994. PMID 32033334
- [Background] Wiegel M, Meston C, Rosen R. The female sexual function index (FSFI): cross-validation and development of clinical cutoff scores. J Sex Marital Ther. 2005 Jan-Feb;31(1):1-20. doi: 10.1080/00926230590475206. PMID 15841702
- [Background] Price DM, Noblett K. Comparison of the cough stress test and 24-h pad test in the assessment of stress urinary incontinence. Int Urogynecol J. 2012 Apr;23(4):429-33. doi: 10.1007/s00192-011-1602-1. Epub 2011 Nov 16. PMID 22086265
- [Background] Guralnick ML, Fritel X, Tarcan T, Espuna-Pons M, Rosier PFWM. ICS Educational Module: Cough stress test in the evaluation of female urinary incontinence: Introducing the ICS-Uniform Cough Stress Test. Neurourol Urodyn. 2018 Jun;37(5):1849-1855. doi: 10.1002/nau.23519. Epub 2018 Jun 21. PMID 29926966
- [Background] Haylen BT, Maher CF, Barber MD, Camargo S, Dandolu V, Digesu A, Goldman HB, Huser M, Milani AL, Moran PA, Schaer GN, Withagen MI. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic organ prolapse (POP). Int Urogynecol J. 2016 Apr;27(4):655-84. doi: 10.1007/s00192-016-3003-y. PMID 26984443
- [Background] González Hinojosa J, Zapico Goñi Á. Diagnóstico médico y tratamientos médico y quirúrgico de las disfunciones del suelo pélvico femenino. Fisioterapia del Suelo Pélvico. Manual para la prevención y el tratamiento en la mujer, en el hombre y en la infancia. Madrid: Editorial Médica Panamericana; 2022. p. 109-25. ISBN: 978-84-9110-453-7.
- [Background] Hall AF, Theofrastous JP, Cundiff GW, Harris RL, Hamilton LF, Swift SE, Bump RC. Interobserver and intraobserver reliability of the proposed International Continence Society, Society of Gynecologic Surgeons, and American Urogynecologic Society pelvic organ prolapse classification system. Am J Obstet Gynecol. 1996 Dec;175(6):1467-70; discussion 1470-1. doi: 10.1016/s0002-9378(96)70091-1. PMID 8987926
- [Background] Navarro Brazalez B, Torres Lacomba M, de la Villa P, Sanchez Sanchez B, Prieto Gomez V, Asunsolo Del Barco A, McLean L. The evaluation of pelvic floor muscle strength in women with pelvic floor dysfunction: A reliability and correlation study. Neurourol Urodyn. 2018 Jan;37(1):269-277. doi: 10.1002/nau.23287. Epub 2017 Apr 28. PMID 28455942
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Vilagut G, Valderas JM, Ferrer M, Garin O, Lopez-Garcia E, Alonso J. [Interpretation of SF-36 and SF-12 questionnaires in Spain: physical and mental components]. Med Clin (Barc). 2008 May 24;130(19):726-35. doi: 10.1157/13121076. Spanish. PMID 18570798
- [Background] Peinado Molina RA, Hernandez Martinez A, Martinez Vazquez S, Martinez Galiano JM. Influence of pelvic floor disorders on quality of life in women. Front Public Health. 2023 Oct 24;11:1180907. doi: 10.3389/fpubh.2023.1180907. eCollection 2023. PMID 37942254
- [Background] Campbell KG, Batt ME, Drummond A. Prevalence of pelvic floor dysfunction in recreational athletes: a cross-sectional survey. Int Urogynecol J. 2023 Oct;34(10):2429-2437. doi: 10.1007/s00192-023-05548-8. Epub 2023 May 10. PMID 37162534
- [Background] Espuna-Pons M, Ros C, Ortega JA, Aliaga F, Perez-Gonzalez A, Palau MJ; Pelvic Floor Research Group (Grup de Recerca del Sol Pelvia, GRESP). Prevalence, incidence, and remission rates of urinary incontinence in women attended in gynecological practice. Neurourol Urodyn. 2017 Apr;36(4):1081-1085. doi: 10.1002/nau.23042. Epub 2016 Jun 6. PMID 27272064
- See also: World Health Organization. Physical Activity — https://www.who.int/es/news-room/fact-sheets/detail/physical-activity
- See also: Spanish Association of Urology. Questionnaires — http://www.aeu.es/cuestionarios.aspx.
- See also: Epidat: epidemiological data analysis' program — https://www.sergas.es/Saude-publica/EPIDAT-4-2